CLINICAL TRIAL: NCT05440266
Title: Electrical Intra-cutaneous Half-sine Stimulation for Optimized Preferential C-fiber Activation in an Established Model of Evoked Pain, Hyperalgesia and Allodynia in Humans (25ms HS Stimulation)
Brief Title: Electrical Intra-cutaneous Half-sine Stimulation for Optimized Preferential C-fiber Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-00682; am22Schneider2
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Pain Perception; Secondary Hyperalgesia
Keywords: C-fiber activation; evoked pain; hyperalgesia; allodynia; half-sine stimulation; 25ms HS stimulation; pain perception; nociceptors; rectangular current stimulation; electrical pain model; numeric rating scale (NRS)
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Intervention Model Description: randomized, crossover, single-blinded experimental proof of concept investigation in healthy volunteers
Who Masked: Participant
Masking Description: Only the study team will know which stimulation will be applied on which intervention. The participant won't be informed about the applied stimulation type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First: half-sine wave stimulation; Second: rectangular shaped stimulation (Active Comparator): First appointment:
  Intracutaneously applied electrical 25 ms half-sine wave stimulation with 2 Hz frequency.
  Second appointment:
  Intracutaneously applied electrical 500 µs rectangular shaped stimulation with 2 Hz frequency.
  Interventions: Diagnostic Test: Study Intervention: 25 ms half-sine wave stimulation; Diagnostic Test: Control Intervention: 500 µs rectangular shaped stimulation
- First: rectangular shaped stimulation; Second: half-sine wave stimulation (Active Comparator): First appointment:
  Intracutaneously applied electrical 500 µs rectangular shaped stimulation with 2 Hz frequency.
  Second appointment:
  Intracutaneously applied electrical 25 ms half-sine wave stimulation with 2 Hz frequency.
  Interventions: Diagnostic Test: Study Intervention: 25 ms half-sine wave stimulation; Diagnostic Test: Control Intervention: 500 µs rectangular shaped stimulation

INTERVENTIONS:
Diagnostic Test: Study Intervention: 25 ms half-sine wave stimulation — Part I: Threshold detection and Flare response: 6 pulses of 25 ms half-sine are given at 2 Hz each, increasing current intensity (mA) until detection threshold, pain threshold and pain level (3 out of 10 NRS) are reached. Determined intensity values reapplied during 214 impulses. Line scan to visualize changes in local skin blood flow done. Part II: Hyperalgesia, Allodynia, Pain and flare response of 65 minutes. Baseline assessment of local skin perfusion and spatial extent of allodynia by using cotton swab and pinprick hyperalgesia. Current intensity is reapplied, adjusted until pain level of 6 reached. After 5 minutes axon reflex flare, allodynia and secondary hyperalgesia are measured and repeated proximal every 10 minutes with last measurement after 65 minutes. In first 15 minutes current intensity is adapted to maintain NRS level of 6. During this 65 minutes' period, 25 ms half-sine is administered continuously.
Diagnostic Test: Control Intervention: 500 µs rectangular shaped stimulation — Part I: Threshold detection and Flare response: 6 pulses of 500 µs rectangular shaped stimulation are given at 2 Hz each, increasing current intensity (mA) until detection threshold, pain threshold and pain level (3 out of 10 NRS) are reached. Determined intensity values reapplied during 214 impulses. Line scan to visualize changes in local skin blood flow done. Part II: Hyperalgesia, Allodynia, Pain and flare response of 65 minutes. Baseline assessment of local skin perfusion and spatial extent of allodynia by using cotton swab and pinprick hyperalgesia. Current intensity is reapplied, adjusted until pain level of 6 reached. After 5 minutes axon reflex flare, allodynia and secondary hyperalgesia are measured and repeated proximal every 10 minutes with last measurement after 65 minutes. In first 15 minutes current intensity is adapted to maintain NRS level of 6. During this 65 minutes' period, 500 µs rectangular shaped stimulation is administered continuously.

SUMMARY:
This exploratory study is to improve an established pain model by a new stimulation profile that allows preferential activation of C fibers that are of main clinical interest in chronic pain and also to generate a stable secondary hyperalgesia, which is of particular interest in the actual research of acute and chronic pain. It is to investigate if the specific activation of afferent sensory fibers and expected lower current intensities makes it more comfortable for the participant as motor neuron activation is much less pronounced at low current intensities. Therefore it compares the area under the curve (AUC) of hyperalgesia during electrical, intracutaneous 25 ms half-sine wave stimulation at a pain level of the numeric rating scale (NRS) of 6 out of 10 for 65 minutes compared to 500 µs rectangular pulses.

DETAILED DESCRIPTION:
Nociceptors in the epidermis are responsible for peripheral pain perception. Mechanical, thermal as well as chemical stimuli can trigger action potentials in nociceptors and thereby pain. Regarding pain, polymodal and "silent" C-fibers are of special interest. Slower depolarisation via sine and half-sine currents preferentially stimulate C-fibers compared to rectangular shaped currents. This study is to compare the development of central sensitization comparing the half-sine wave and the rectangular stimulation, hypothesizing that preferential C fiber stimulation through half-sine currents facilitate the development of secondary hyperalgesia.

This exploratory study is to improve an established pain model by a new stimulation profile that allows preferential activation of C fibers that are of main clinical interest in chronic pain and also to generate a stable secondary hyperalgesia, which is of particular interest in the actual research of acute and chronic pain. It is to investigate if the specific activation of afferent sensory fibers and expected lower current intensities makes it more comfortable for the participant as motor neuron activation is much less pronounced at low current intensities. Therefore it compares the area under the curve (AUC) of hyperalgesia during electrical, intracutaneous 25 ms half-sine wave stimulation at a pain level of the numeric rating scale (NRS) of 6 out of 10 for 65 minutes compared to 500 µs rectangular pulses.

Every volunteer will have two appointments. There will be a "washout" period of at least two weeks between the two appointments. On each day two microdialysis catheters containing internally a stainless steel wire will be inserted intracutaneously on the volar surface of the adominant forearm for a length of approximately 10 mm and at a distance of 5 mm. Before insertion, the catheters are filled with 0.9% saline and after insertion a continuous flow of 0.4 μl/min will be ensured by a syringe pump (Perfusor®) to facilitate conduction and to protect the tissue from potential local pH changes by the direct current. Alternating polarity of the both pulses is used to ensure charge-balanced stimulation.

It is randomly assigned which current form is applied on the first and on the second trial. Subsequently, the stainless steel wire serving as electrodes of the current generator (for 25 ms half-sine stimulation the Digitimer DS5; Digitimer Ltd, Hertfordshire, United Kingdom; and for 500 µs rectangular stimulation the Digitimer DS7A; Digitimer Ltd, Hertfordshire, United Kingdom) are connected. The rectangular pulses are generated by the Digitimer DS7A, which works in combination with a pulse generator (PG 1, Rimkus Medizintechnik, Parsdorf, Germany)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (18 - 65 years old, American Society of Anaesthesiologists (ASA) I or II)
* BMI between 18.5 until 25 kg/m2
* Able to understand the study and the NRS scale
* Able to give informed consent

Exclusion Criteria:

* Regular intake of medications or drugs potentially interfering with pain sensation (analgesics, opioids, antihistamines, calcium and potassium channel blockers, serotonin / noradrenaline reuptake inhibitors, corticosteroids)
* Neuropathy
* Chronic pain
* Neuromuscular disease
* Dermatological disease as Atopic Dermatitis
* Psychiatric disease
* Pregnancy / Lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Secondary hyperalgesia measured by the area under the curve (AUCHyperHS) | 65 minutes from start of stimulation until stop of stimulation
  Difference between the AUC of secondary hyperalgesia during 25ms half-sine wave stimulation (AUCHyperHS) at pain level NRS 6 for 65 minutes and the AUC of secondary hyperalgesia measured during 500µs rectangular shaped stimulation (AUCHyperRect) at pain level NRS 6 for 65 minutes

SECONDARY OUTCOMES:
Number of pulses needed to reach 25% of the final extent of the flare response | approx. 65 minutes at each intervention day (first appointment and second appointment)
  The number of pulses needed to reach 25% of the final extent of the flare response (measured with a laser Doppler line scan while applying 214 impulses in total) at detection and pain threshold and at pain level NRS 3.
Needed time (in minutes) to generate 50% of the final extent of secondary hyperalgesia. | approx. 65 minutes at each intervention (first appointment and second appointment)
  Difference between the needed time (in minutes) to generate 50% of the final extent of secondary hyperalgesia during 25ms half-sine wave stimulation and during 500µs rectangular shaped stimulation.
Current intensity needed to reach same pain level (NRS 6) | approx. 65 minutes at each intervention day (first appointment and second appointment)
  Difference of the amount of current intensity needed to reach same pain level (NRS 6) after adaption during the first 15 minutes of stimulation between half-sine and rectangular currents (0 = no pain and 10 = maximum tolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Schneider, Dr. med., Principal Investigator — Department of Anaesthesiology, University Hospital of Basel (USB)
Locations (1):
- Department of Anaesthesiology, University Hospital of Basel (USB), Basel, Switzerland